CLINICAL TRIAL: NCT01003509
Title: A New Approach in Inguinal Hernia Repair: Double Repair. A Prospective, Randomized, Controlled Clinical Trial
Acronym: herni
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: No any sponsor, No any sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hernia; aysan (Other: Bezmialem vakif University)
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Hernia
Keywords: inguinal; hernia; new; repair; modified shouldice; double
MeSH Terms: conditions — Hernia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study, control (No Intervention): Control: Only modified shouldice repair performed Study: Modified Shouldice + Moloney repairs performed
- modified shouldice and double (No Intervention): one arm is only modified shouldice, other one is double
  Interventions: Procedure: modified shouldice and double

INTERVENTIONS:
Procedure: modified shouldice and double — one arm modified shouldice, other one is double repair
  Other Names: control group, study group
  Arms: modified shouldice and double

SUMMARY:
This is a new inguinal hernia repair technique.

DETAILED DESCRIPTION:
In this study we are revealing a new inguinal hernia repair technique. It is constructed from two layers. Deep layer is modified Shouldice technique, the other superficial one is moloney technique.

ELIGIBILITY:
Inclusion Criteria:

* Inguinal hernia

Exclusion Criteria:

* Recurrences, child

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-01; Primary Completion 2006-01 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
complications, recurrences | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Arslan Kaygusuz, surgeon, Study Chair — S.B. Istanbul Educational & Teaching Hospital
Locations (1):
- S.B. Istanbul Educational & Teaching Hospital, Istanbul, Marmara, Turkey (Türkiye)